CLINICAL TRIAL: NCT06575855
Title: Comparative Effectiveness of Instrument Assisted Soft Tissue Mobilization IASTM and Muscle Energy Technique MET on Post Operative Elbow Stiffness
Brief Title: Comparative Effectivenes of IASTM and MET on Post Operative Elbow Stiffness
Acronym: IASTM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Faisalabad (Other)
Collaborators: University of Sargodha (Other)
Responsible Party: Principal Investigator, Nayyab Goher, Student, University of Faisalabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: nayyabgoher999@gmail.com
Record Dates: First submitted 2024-08-23; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Elbow Stiffness
Keywords: Post operative elbow stiffness, MET, IASTM

STUDY DESIGN:
Intervention Model Description: 28 participants divided in to two groups, Group A and Group B
Masking Description: Patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Group A received IASTM as treatment protocol
  Interventions: Other: IASTM
- Group B (Active Comparator): Group B received METs as a treatment protocol
  Interventions: Other: METS

INTERVENTIONS:
Other: IASTM — Group A received IASTM by using Graston Tool
  Arms: Group A
Other: METS — Group B received METs
  Arms: Group B

SUMMARY:
This study is basically for the evaluation of comparative effectiveness of instrument assisted soft tissue mobilization IASTM and muscle energy technique MET on Post operative , Randomized clinical trial .

DETAILED DESCRIPTION:
In this study 28 participants including, which is further devided into two groups,14 in each group which is named as Group A,and Group B respectively.these groups are randomly allocated and give them intervention.which is instrument assisted soft tissue mobilization IASTM given to Group A and muscle energy technique MET given to Group B,then compare the effectiveness of both groups on Post operative elbow stiffness, duration of protocol is basically for 2,3 weeks depending upon patient condition and present situation.

ELIGIBILITY:
Inclusion Criteria:

* gender both Age:30 to 50 years Who fullfil concent form

Exclusion Criteria:

* other than inclusion criteria

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 28 (Actual)
Dates: Start 2024-02-17 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
VAS and goniometer | 4 months
  Visual analog scaleThe Visual Analog Scale (VAS) is a 10 cm line with anchor statements on the left (no pain) and on the right (extreme pain) and universal goniometer to measure the range of motion, an instrument that measures angle motion at a joint.

SECONDARY OUTCOMES:
DASH questionaire | 4 months
  The disabilities of the arm, shoulder and hand (DASH) questionnaire is a self-administered region-specific outcome instrument developed as a measure of self-rated upper-extremity disability and symptoms. The DASH consists mainly of a 30-item disability/symptom scale, scored 0 (no disability) to 100

CONTACTS AND LOCATIONS:
Locations (1):
- Nayyab Goher, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No